CLINICAL TRIAL: NCT04924218
Title: The Effect of Endoscopic Procedures After Radical Prostatectomy on Urinary Incontinence
Brief Title: Evaluation of the Effect of Endoscopic Urethral Procedures Applied After Radical Prostatectomy on Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, selman unal, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AnkaraYBU-URO-SU-01
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer; Incontinence
Keywords: Prostate Cancer; Urinary Incontinence; Endoscopic Surgical Procedures
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rigid cystoscopy (Active Comparator): Group undergoing endoscopic urethral procedure with rigid cystoscopy after radical prostatectomy
  Interventions: Procedure: endoscopic surgical intervention
- flexible cystoscopy (Active Comparator): Group undergoing endoscopic urethral procedure with flexible cystoscopy after radical prostatectomy
  Interventions: Procedure: endoscopic surgical intervention
- semi-rigid ureterorenoscopy (Active Comparator): Group undergoing endoscopic urethral procedure with semi-rigid ureterorenoscopy after radical prostatectomy
  Interventions: Procedure: endoscopic surgical intervention

INTERVENTIONS:
Procedure: endoscopic surgical intervention — The researchers investigated whether endoscopic surgical procedures performed due to various indications (hematuria, urinary tract stone, suspected bladder mass) in the patient group who had undergone radical prostatectomy, caused a change in urinary incontinence level. The researchers divided the endoscopic instruments used into 3 groups and evaluated whether there was a difference in urinary incontinence level between rigid cystoscope, flexible cystoscope and ureterorenoscope groups.

SUMMARY:
The researchers investigated whether endoscopic retrograde urethral interventions applied for various reasons after radical prostatectomy (RP) operation cause a change in urinary incontinence (UI) level, and if there is a change, whether it changes according to the endoscopic procedure time and the endoscopic instrument used.

DETAILED DESCRIPTION:
Localized prostate cancer is usually treated with RP. The most common complications after RP are erectile dysfunction (ED) and UI. After RP, some patients may require retrograde endoscopic urethral intervention. In this study, researchers investigated whether there is a change in the UI level in patients that underwent retrograde urethral intervention after RP and whether this change was affected by the duration of the procedure and type of endoscopic device used.

Methods: Eighteen patients were included in the study. The patients were divided into 3 groups based on the endoscopic device used: group 1 rigid cystoscopy, group 2 flexible cystoscopy, and group 3 semi-rigid ureterorenoscopy (URS). The Turkish version of the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) and the number of pads used daily was questioned before the endoscopic procedure and 1 month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone radical prostatectomy
* Patients that had undergone an endoscopic procedure 1 year after RP

Exclusion Criteria:

* Patients with urinary tract infection before the endoscopic procedure,
* Urinary tract infection at 1st month follow-up
* Central neurological deficit
* History of adjuvant radiotherapy after RP
* Bladder neck stenosis and urethral stenosis
* Patients that had undergone endoscopic urethral intervention before this scheduled procedure
* Patients who had a double J stent inserted during the endoscopic procedure and required a second endoscopic intervention
* Patients that required the use of bipolar or monopolar cautery

Ages: 52 Years to 84 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) | 1 month
  The ICIQ-UI Short Form is a questionnaire for evaluating the frequency, severity and impact on quality of life (QoL) of urinary incontinence in men and women in research and clinical practice across the world. Minimum score: 0, maximum score: 21. The higher the score, the higher the level of urinary incontinence is interpreted.
Daily pad use | 1 month
  It refers to the number of pads used in 1 day due to urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Onder Kayigil, Professor, Study Chair — Ankara Yildirim Beyazit University School of Medicine
Locations (1):
- Ankara Yildirim Beyazit University, Schhol of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No